CLINICAL TRIAL: NCT03924362
Title: A Prospective Trial of Feasibility and Efficacy of Simultaneous Bilateral Percutaneous Nephrolithotomy
Brief Title: Bilateral Percutaneous Nephrolithomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ben Chew, MD, Associate Professor, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H19-00426
Record Dates: First submitted 2019-03-26; First posted 2019-04-23 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Nephrolithiasis of Both Kidneys

STUDY DESIGN:
Intervention Model Description: Patients will be managed either with simultaneous bilateral procedures or staged unilateral procedures based on surgeon's routine practice pattern. Additional surgical interventional will be dependent on initial patient stone-free outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simultaneous Bilateral PCNL (Active Comparator): Patients undergo simultaneous bilateral PCNL.
  Interventions: Procedure: PCNL
- Unilateral PCNL (Active Comparator): Patients undergoing unilateral staged PCNL.
  Interventions: Procedure: PCNL

INTERVENTIONS:
Procedure: PCNL — Percutaneous Nephrolithotomy is a means of treating large kidney stone burdens.

SUMMARY:
The purpose of this study is to determine the effective regimen for definitive surgical therapy of bilateral kidney stones. It is unknown whether patients who undergo simultaneous bilateral percutaneous nephrolithotomy (PCNL) experience improved post-operative outcomes compared to patients who have staged unilateral procedures.

DETAILED DESCRIPTION:
Purpose:

The aim of this research is to determine an effective regimen for definitive surgical therapy of bilateral kidney stones. It is unknown whether patients who undergo simultaneous bilateral percutaneous nephrolithotomy (PCNL) experience improved post-operative outcomes compared to patients who have staged unilateral procedures.

Hypothesis and Justification The gold standard for surgical management of large kidney stones is percutaneous nephrolithotomy (PCNL). A large renal stone burden has been defined as >20mm. In addition, PCNL has improved stone-free rates for lower pole calculi >10mm compared to alternative treatments. Guidelines encourage removal of staghorn calculi for surgical candidates (Assimos et al., 2016). Patients with bilateral large stone burdens have been managed with one of two general options: (i) a single procedure in which both kidneys are operated upon or (ii) two separate procedures in which only one kidney is addressed per procedure. However, there are no prospectively performed peer-reviewed studies directly comparing the two practices. The investigators seek to determine whether there is a significant difference in patient outcomes based on the surgical regimen chosen.

The investigators hypothesize that in comparison to unilateral PCNL (U-PCNL), simultaneous bilateral PCNL (SB-PCNL) under one anesthetic results in comparable

1. stone free rates
2. re-intervention rates for residual stones and
3. perioperative complication rates

Objectives

The objectives are:

1. To provide clinical data on outcomes following simultaneous bilateral and staged percutaneous nephrolithotomy for renal and ureteral calculi
2. To determine patient preference with respect to simultaneous versus staged PCNL

Research Design This study will be a prospective, non-randomized, multi-centre, non-blinded trial. Participants will be accrued through the Vancouver General Hospital Stone Center who have been referred for bilateral stones or have been seen in consultation for bilateral stones at the Department of Urologic Sciences and are scheduled for a percutaneous nephrolithotomy (PCNL). Consent forms and Letters of Introduction outlining the study will be given to patients by a research coordinator once the decision is made to book surgery. Patients will have at least 24 hours to decide to participate. Patients will receive surgical management for their stones in the form of PCNL. A computed tomography (CT) scan of the kidneys will be performed post-operatively by week 6 to determine if any residual stone fragments are present. Patients will be seen in follow up at 3 months in clinic after undergoing a follow up CT KUB, renal ultrasound, or KUB as necessary to evaluate stone clearance.

ELIGIBILITY:
Inclusion Criteria:

All subjects with a clinical diagnosis of struvite calculi will potentially be included. Specific inclusion criteria include the following:

1. Age >18 years
2. Any patient with bilateral stone burden eligible and appropriate for PCNL procedure
3. Medically fit for definitive surgical management of stone.

Exclusion Criteria:

Patients with any of the following characteristics will not be eligible for the present study:

1. Those with medical comorbidities preventing them from safely undergoing definitive surgical therapy.
2. Patients who are unable to provide informed consent.
3. Patients who are planned for alternative procedures (ureteroscopy, extracorporeal shock wave lithotripsy)
4. Anyone who is unable to give their informed consent
5. Anyone under the age of 19
6. Anyone who, in the opinion of the PI, is unfit or unsuitable to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Stone Free Rates Measured using Chi-Square analysis. | 3 months.
  Rate of clearance of kidney stones following the procedure.
Number of Participants with Repeat procedures | 3 months.
  Number of Participants requiring repeat surgical procedures for residual stones following initial treatment.

SECONDARY OUTCOMES:
Length of hospital stay | 3 months.
  Hospital stay for simultaneous bilateral versus staged PCNL.
Number of Participants with Complications | 3 months.
  Number of participants with perioperative complication and rates for each procedure.
Patient Quality of Life | 3 months.
  Quality of life assessment comparing the two different procedures will be conducted with the Wisconsin Stone Quality of Life questionnaire (WISQOL). WISQOL is a disease-specific, health-related quality of life measure designed for patients who form kidney stones. This questionnaire has 4 different domains: social-domain 1, emotional-domain 2, stone related-domain 3 and vitality-domain 4. In the questionnaire, patients are to answer between 1 (Very true) to 5 (Not true at all). 1 is the worst outcome, and 5 is the best outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Chew, MD, Principal Investigator — University of British Columbia, Associate Professor
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
The University of British Columbia is the main site of the study, therefore all data will be transferred from the subsites to the University of British Columbia, and no transfer of data to the subsites. Any data transfer will be de-identified.

REFERENCES:
- [Background] Assimos D, Krambeck A, Miller NL, Monga M, Murad MH, Nelson CP, Pace KT, Pais VM Jr, Pearle MS, Preminger GM, Razvi H, Shah O, Matlaga BR. Surgical Management of Stones: American Urological Association/Endourological Society Guideline, PART II. J Urol. 2016 Oct;196(4):1161-9. doi: 10.1016/j.juro.2016.05.091. Epub 2016 May 27. PMID 27238615
- [Background] Jones P, Dhliwayo B, Rai BP, Mokete M, Amitharaj R, Aboumarzouk OM, Somani BK. Safety, Feasibility, and Efficacy of Bilateral Synchronous Percutaneous Nephrolithotomy for Bilateral Stone Disease: Evidence from a Systematic Review. J Endourol. 2017 Apr;31(4):334-340. doi: 10.1089/end.2016.0851. Epub 2017 Mar 22. PMID 28326800
- [Background] Kang SK, Cho KS, Kang DH, Jung HD, Kwon JK, Lee JY. Systematic review and meta-analysis to compare success rates of retrograde intrarenal surgery versus percutaneous nephrolithotomy for renal stones >2 cm: An update. Medicine (Baltimore). 2017 Dec;96(49):e9119. doi: 10.1097/MD.0000000000009119. PMID 29245347
- [Background] Penniston KL, Antonelli JA, Viprakasit DP, Averch TD, Sivalingam S, Sur RL, Pais VM Jr, Chew BH, Bird VG, Nakada SY. Validation and Reliability of the Wisconsin Stone Quality of Life Questionnaire. J Urol. 2017 May;197(5):1280-1288. doi: 10.1016/j.juro.2016.11.097. Epub 2016 Nov 23. PMID 27889419
- [Background] Silverstein AD, Terranova SA, Auge BK, Weizer AZ, Delvecchio FC, Pietrow PK, Munver R, Albala DM, Preminger GM. Bilateral renal calculi: assessment of staged v synchronous percutaneous nephrolithotomy. J Endourol. 2004 Mar;18(2):145-51. doi: 10.1089/089277904322959770. PMID 15072621
- [Background] Wang CJ, Chang CH, Huang SW. Simultaneous bilateral tubeless percutaneous nephrolithotomy of staghorn stones: a prospective randomized controlled study. Urol Res. 2011 Aug;39(4):289-94. doi: 10.1007/s00240-010-0342-x. Epub 2010 Dec 16. PMID 21161650